CLINICAL TRIAL: NCT03444259
Title: Cardiovascular Research Consortium - a Prospective Project to Identify Biomarkers of Morbidity and Mortality in Cardiovascular Interventional Patients
Brief Title: Prospective Project to Identify Biomarkers of Morbidity and Mortality in Cardiovascular Interventional Patients
Acronym: CAREBANK
Status: Active, not recruiting | Type: Observational
Sponsor: University of Turku (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Tuomas Kiviniemi, Cardiologist, MD, PhD, FESC, University of Turku
Other Study IDs: T273/2015
Record Dates: First submitted 2018-02-15; First posted 2018-02-23 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation; Coronary Artery Disease; Aortic Valve Stenosis; Aortic Valve Disease; Mitral Valve Disease; Cardiac Arrythmias; Cardiac Tumor; Cardiac Surgery
Keywords: Atrial fibrillation; Aortic stenosis; Coronary artery disease; Cardiac surgery; Atrial appendage
MeSH Terms: conditions — Atrial Fibrillation; Coronary Artery Disease; Aortic Valve Stenosis; Aortic Valve Disease; Heart Neoplasms | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Atrial appendage, valves, ascending aorta, pericardium
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Atrial fibrillation: Patients with atrial fibrillation
  Interventions: Procedure: Cardiac surgery
- Coronary bypass: Patients undergoing coronary bypass
  Interventions: Procedure: Cardiac surgery
- Aortic valve replacement: Patients undergoing aortic valve replacement
  Interventions: Procedure: Cardiac surgery
- Mitral valve repair: Patients undergoing mitral valve repair
  Interventions: Procedure: Cardiac surgery
- Other: Patients undergoing cardiac surgery for indication other than above
  Interventions: Procedure: Cardiac surgery

INTERVENTIONS:
Procedure: Cardiac surgery — Open heart surgery

SUMMARY:
The objective of CAREBANK study is to establish definitive relationships with human cardiac samples and clinical phenotypes in patients undergoing cardiac procedures. Specifically, the investigators aim at comparing atrial phenotypes from atrial fibrillation patients and controls. The work consists of three broad categories: A) role of atrial cardiomyopathy in atrial fibrillation; B) genetic defects predisposing to atrial fibrillation; and C) the role of inflammation in atrial fibrillation.

DETAILED DESCRIPTION:
The investigators aim to A) compare atrial cardiomyopathy findings from the tissue samples to clinical phenotype and adverse events B) study the association of genetic defects predisposing to atrial fibrillation with atrial cardiomyopathy findings in the tissue samples C) assess the role of inflammation in atrial fibrillation by comparing circulating cytokine profiles, purinergic signaling and atrial cardiomyopathy findings in tissue samples.

ELIGIBILITY:
Inclusion Criteria:

* Any open-heart cardiac surgery
* Written informed consent
* All-comers design

Exclusion Criteria:

* No informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing open-heart cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 1001 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation | postoperatively until 5 years follow-up
  Occurrence of atrial fibrillation

SECONDARY OUTCOMES:
Stroke | postoperatively until 5 years follow-up
  Occurrence of stroke
Transient ischemic attack | postoperatively until 5 years follow-up
  Occurrence of Transient ischemic attack
Myocardial infarction | postoperatively until 5 years follow-up
  Occurrence of Myocardial infarction
Target vessel revascularization | postoperatively until 5 years follow-up
  Occurrence of Target vessel revascularization
All-cause Mortality | postoperatively until 5 years follow-up
  All-cause Mortality
Post-pericardiotomy syndrome | postoperatively until 1 years follow-up
  Occurrence of Post-pericardiotomy syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Tuomas O Kiviniemi, MD, PhD, Study Director — Turku University Hospital; Jarmo Gunn, MD, PhD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Maaniitty E, Sinisilta S, Jalkanen J, Vasankari T, Biancari F, Gunn J, Jalkanen S, Airaksinen KEJ, Hollmen M, Kiviniemi T. Distinct circulating cytokine levels in patients with angiography-proven coronary artery disease compared to disease-free controls. Int J Cardiol Cardiovasc Risk Prev. 2024 Jul 4;22:200307. doi: 10.1016/j.ijcrp.2024.200307. eCollection 2024 Sep. PMID 39091640
- [Derived] Maaniitty E, Jalkanen J, Sinisilta S, Gunn J, Vasankari T, Biancari F, Jalkanen S, Airaksinen KEJ, Hollmen M, Kiviniemi T. Differential circulating cytokine profiles in acute coronary syndrome versus stable coronary artery disease. Sci Rep. 2024 Jul 27;14(1):17269. doi: 10.1038/s41598-024-68333-7. PMID 39068298
- [Derived] Viikinkoski E, Jalkanen J, Gunn J, Vasankari T, Lehto J, Valtonen M, Biancari F, Jalkanen S, Airaksinen KEJ, Hollmen M, Kiviniemi TO. Red blood cell transfusion induces abnormal HIF-1alpha response to cytokine storm after adult cardiac surgery. Sci Rep. 2021 Nov 15;11(1):22230. doi: 10.1038/s41598-021-01695-4. PMID 34782683